CLINICAL TRIAL: NCT06460597
Title: Comparative Effects of Papworth Technique Versus Pranayama in Asthmatic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0382
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Asthma
Keywords: asthma,; Anxiety,; Papworth Technique
MeSH Terms: conditions — Asthma; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papworth Technique (Experimental): The Papworth breathing technique is used by respiratory physiotherapists to control and correct breathing. Instead of using the chest, Papworth technique encourages to take more relaxed breathing by using the abdomen. Breathing in slowly through the nose and breathing out through pursed lips as if blowing out a candle. Repeat this cycle for 3-5 times
  Interventions: Other: Papworth Technique
- Pranayama (Active Comparator): Pranayama is an ancient breath technique that originates from yogic practices in India. Sitting comfortably, slowly inhale through the nose and count to five. Direct the breath across the back of the throat as you inhale so the air makes a slight hissing sound keeping the lips sealed, breathe out through the nose and try to match the length of your inhale. The breath should make a noise like waves crashing as you exhale. Continue to inhale and exhale using the same process for 5 to 8 minutes. Aim to do this exercise for 10 to 15 minutes as become more practiced.
  Interventions: Other: Pranayama

INTERVENTIONS:
Other: Papworth Technique — The Papworth breathing technique is used by respiratory physiotherapists to control and correct breathing. Instead of using the chest, Papworth technique encourages to take more relaxed breathing by using the abdomen. Breathing in slowly through the nose and breathing out through pursed lips as if blowing out a candle. Repeat this cycle for 3-5 times
  Arms: Papworth Technique
Other: Pranayama — Pranayama is an ancient breath technique that originates from yogic practices in India. Sitting comfortably, slowly inhale through the nose and count to five. Direct the breath across the back of the throat as you inhale so the air makes a slight hissing sound keeping the lips sealed, breathe out through the nose and try to match the length of your inhale. The breath should make a noise like waves crashing as you exhale. Continue to inhale and exhale using the same process for 5 to 8 minutes. Aim to do this exercise for 10 to 15 minutes as become more practiced.
  Arms: Pranayama

SUMMARY:
Asthma is a chronic and heterogeneous disease characterized by reversible airway obstruction, airway inflammation and bronchial damage causing dyspnea, wheezing, chest tightness, coughing and impaired quality of life. Papworth technique and Pranayama modify the pattern of breathing to reduce the hyperventilation resulting in normalization of CO2 levels, reduction of bronchospasm and resulting breathlessness

.These techniques also change the emotional stresses, improve the immunity system and improve the strength /endurance of respiratory muscles. After taking the consent form from the participants, data will be collected from Gulab Devi Chest Hospital. Non-Probability Convenience Sampling will be applied on asthmatic patients according to inclusion criteria. Patients will be allocated through simple random sampling into group A and B to collect data. Group A will be treated by Papworth technique. Four weeks will be required to complete the treatment plan. Three sessions will be given for one week so total 12 sessions will be given in one month. Group B will be treated by Pranayama. Four weeks will be required to complete the treatment plan. Three sessions will be given for one week so total 12 sessions will be given in one month. Papworth Technique and Pranayama are used and are assessed to see their effectiveness in asthmatic patients by using four questionnaires on dyspnea, fatigue, anxiety, depression and quality of life. These four standardized questionnaires are Borg Dyspnea Scale (BDS), Modified Fatigue Impact Scale (MFIS), Hospital Anxiety Depression Scale (HADS) and Asthma Quality of life. Pulse oximeter will be used to check the oxygen saturation. The study duration will be completed within time duration of 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Both genders(male and female)
* Age 20-40 years
* Patients with adverse mood effects
* Mild to moderate chronic asthma

Exclusion Criteria:

* Acute severe asthma
* Chronic chest infections like TB
* Chest deformity
* Bronchiectasis
* Cardiac Disease
* Substance abusers
* Chronic Obstructive Pulmonary Disease
* Neurological Disorders

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Pulse Oximeter | baseline and fourth week
  oxygen saturation
Hospital Anxiety Depression Scale | baseline and fourth week
  It is a self- assessment scale. It is a reliable instrument for detecting the anxiety and depression in patients with asthma. The anxiety and depressive subscales are also valid measures of severity of emotional stresses. The HADS is a self-report rating scale consists of 14 items on a 4 point Likert Scale range from 0-3.It measures anxiety and depression, 7 items for each subscale. The total score is the sum of 14 items and for each subscale is the sum of respective seven items, ranging from 0-21
Asthma Quality of life | baseline and fourth week
  It has 32 questions that contains four sub domains, these are symptoms 11 items, activity limitations 12, emotional function 5, environmental stimuli 4 items. This is marked on a 7 point Likert scale that is changing from 1 to 7 where higher scores indicate better quality of life,1 indicates severely impaired patients with asthma while 7 indicates no impairments. Asthma quality of life has strong measurement properties and is valid for measuring health related quality of life in asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Chest Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sockrider M, Fussner L. What Is Asthma? Am J Respir Crit Care Med. 2020 Nov 1;202(9):P25-P26. doi: 10.1164/rccm.2029P25. No abstract available. PMID 33124914
- [Background] Gans MD, Gavrilova T. Understanding the immunology of asthma: Pathophysiology, biomarkers, and treatments for asthma endotypes. Paediatr Respir Rev. 2020 Nov;36:118-127. doi: 10.1016/j.prrv.2019.08.002. Epub 2019 Oct 9. PMID 31678040
- [Background] Miller RL, Grayson MH, Strothman K. Advances in asthma: New understandings of asthma's natural history, risk factors, underlying mechanisms, and clinical management. J Allergy Clin Immunol. 2021 Dec;148(6):1430-1441. doi: 10.1016/j.jaci.2021.10.001. Epub 2021 Oct 14. PMID 34655640